CLINICAL TRIAL: NCT05657834
Title: A Phase I, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-TVB-2640 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Open-label Study of the Absorption, Metabolism, and Excretion of [14C]TVB-2640 Following a Single Oral Dose in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SB2640-CLIN-008
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers
Keywords: Absorption; Metabolism; Excretion; Radiolabeled Dose; Mass Balance [14C]

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm 1 (Experimental): Single dose of TVB-2640, 50 mg, oral administration
  Interventions: Drug: [14C]-TVB-2640

INTERVENTIONS:
Drug: [14C]-TVB-2640 — 50 mg of TVB-2640 oral administration

SUMMARY:
A Phase 1, Open-label Study of the absorption, metabolism, and excretion of a single oral dose of [14C]TVB-2640 healthy male subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Males, of any race, between 19 and 55 years of age, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and Check-in as assessed by the Investigator (or designee).
* History of a minimum of 1 bowel movement per day

Key Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of corneal edema, keratitis, xerophthalmia (dry eye), or other corneal abnormalities.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (cholecystectomy will not be allowed; uncomplicated appendectomy and hernia repair will be allowed).
* Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines.
* Use of any sensitive substrates of cytochrome P450 (CYP)2C9 or CYP3A4/5, or inhibitors of CYP3A4 within 30 days prior to IMP administration (Day 1).
* Donation or loss of ≥ 550 mL blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
[14C]TVB-2640: AUC-inf in plasma | Up to 22 days
[14C]TVB-2640: Amount excreted in urine | Up to 22 days
[14C]TVB-2640: Amount excreted in feces | Up to 22 days

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No